CLINICAL TRIAL: NCT00357721
Title: Randomized, Open-Label, Multiple-Dose Study to Evaluate the Pharmacokinetics of Atazanavir Administered Twice-Daily in Health Subjects
Brief Title: Atazanavir Twice Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AI424-286
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections; Protease Inhibitor
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

ARMS (3):
- A1 (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate
- A2 (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate
- A3 (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate

INTERVENTIONS:
Drug: Atazanavir Sulphate — Capsules, Oral, 200 mg, twice daily, 7 days.
  Other Names: Reyataz
  Arms: A1
Drug: Atazanavir Sulphate — Capsules, Oral, 300 mg, twice daily, 8 days.
  Other Names: Reyataz
  Arms: A2
Drug: Atazanavir Sulphate — Capsules, Oral, 400 mg, twice daily, 9 days.
  Other Names: Reyataz
  Arms: A3

SUMMARY:
The purpose of this clinical research study is to assess the pharmacokinetics of atazanavir administered twice-daily relative to historical data from atazanavir/ritonavir 300/100 mg, given once daily.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 to 45 years old with a BMI of 18 to 30 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Assess the pharmacokinetics (PK) of atazanavir administered twice-daily (BID) relative to historical data from atazanavir/ritonavir 300/100 mg, given once-daily.

SECONDARY OUTCOMES:
Assess the dose proportionality and the diurnal variation in the PK of atazanavir given BID
Assess the effect of atazanavir BID on bilirubin values and explore the relationship between bilirubin and atazanavir dose level/exposure by UGT1A1 genetic isoform
Assess the effect of atazanavir BID on metabolic parameters
Assess the safety and tolerability of atazanavir when administered BID

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States